CLINICAL TRIAL: NCT00540891
Title: The Efficacy, Onset of Effect, and Safety of Alfuzosin Once Daily in the Treatment of Lower Urinary Tract Symptoms of Benign Prostatic Hyperplasia: A Randomized, Placebo-Controlled Trial Using an Acute International Prostate Score
Acronym: ALF-ACUTE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L_8472
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Last update posted 2007-10-08 (Estimated); Status verified 2007-10

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — alfuzosin

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: ALFUZOSIN

SUMMARY:
Primary: Evaluate the safety and onset of symptom relief using an acute I-PSS form (7 day form).

Determine onset of urinary peak flow improvement after 7 days Secondary: Determine improvement in Bother Score after 7 & 28 days; improvement in sexual function after 28 days; assess one-month efficacy and safety

ELIGIBILITY:
Inclusion Criteria:

- Men aged greater than or equal to 50 years with a history of lower urinary tract symptoms (LUTS) related to BPH for greater than or equal to 6 months, an International Prostate Symptom Score (I-PSS) (0 to 35 points scale) of at least 13 points, a maximum urinary flow rate (Qmax) between 5 and 12 mL/sec (with a voided volume of greater than or equal to 150 mL), a residual urine volume of less than or equal to 350 mL, and a bothersomeness score (0 to 6 points scale) of at least 3 points. All patients will undergo prostate size assessment by transrectal ultrasonography (TRUS) if not done within past 12 months.

Exclusion Criteria:

- Include, but are not limited to: concomitant lower urinary tract disease; previous prostatic surgery; history of postural hypotension or syncope; concomitant use of medications that may alter the voiding pattern; and clinically relevant biochemical abnormalities. Patients with a serum prostate-specific antigen (PSA) >10 ng/mL will be excluded, and those with an elevated serum PSA between 4 and 10 ng/mL must have prostate cancer excluded to the satisfaction of the investigator.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2003-02; Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and onset of symptom relief using an acute I-PSS form(7 day form). | 7 day
Determine onset of urinary peak flow improvement | after 7 days

SECONDARY OUTCOMES:
Determine improvement in Bother Score | after 7 & 28 days
To determine the improvement in sexual function | after 28 days
Assess one-month efficacy and safety | one month

CONTACTS AND LOCATIONS:
Overall Officials: Yasir Nagarwala, M.D., Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States